CLINICAL TRIAL: NCT05533203
Title: A Multicenter, Non-randomized, Open-label, and Dose-escalation Phase I Study to Evaluate the Safety of Prodencel Treatment in Patients With Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Safety of Prodencel in the Treatment of Metastatic Castration-resistant Prostate Cancer (mCRPC)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Humantech Biotechnology Co. Ltd (Industry)
Collaborators: Shanghai Changhai Hospital,The First Affiliated Hospital of Naval Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTB-B003-I
Record Dates: First submitted 2022-09-01; First posted 2022-09-08 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: metastatic castration-resistant prostate cancer; dendritic cell vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prodencel Treated for mCRPC (Experimental): Cohort 1: Each subject would receive Prodencel treatment at a dose of 5×10^6 cells every two weeks for a total of 3 doses.
  Cohort 2: Each subject would receive Prodencel treatment at a dose of 10×10^6 cells every two weeks for a total of 3 doses.
  Cohort 3: Each subject would receive Prodencel treatment at a dose of 15×10^6 cells every two weeks for a total of 3 doses.
  Cohort 4: The safe and effective dose from cohort 1-3 is recommended for booster immunization of cohort 4. Subjects will receive additional Prodencel treatment every 4 weeks, until disease progression or intolerance after the 3 doses of immune induction, to evaluate the safety and tolerability of the booster immunization.
  Interventions: Biological: Prodencel; an autologous dendritic cell therapeutic tumor vaccine

INTERVENTIONS:
Biological: Prodencel; an autologous dendritic cell therapeutic tumor vaccine — Subcutaneous injection, each injection point should not exceed 1ml.

SUMMARY:
This phase I clinical trial is to evaluate the safety of Prodencel (an autologous dendritic cell therapeutic tumor vaccine.) in patients with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This is a single arm pilot study to evaluate the safety of delivering a dendritic cell vaccine in fifteen to twenty-four (n=15-24) adult patients diagnosed with prostate adenocarcinoma after novel androgen-deprived therapy and docetaxel chemotherapy failure. The study is constructed in a 3+3 design for three steps of dose escalation with rigorous and mandatory safety monitoring. Subjects received the vaccine at a dose of 5-15×10^6 cells every two weeks for a total of 3 doses. A dose from cohort 1-3 is recommended for booster immunization every 4 weeks until disease progression or intolerance, to evaluate the safety and tolerability of the booster immunization of Prodencel. Subjects will be monitored for adverse events as dictated by CTCAE version 5.

ELIGIBILITY:
Inclusion Criteria：

* Histologically prostate adenocarcinoma, exclusion of the initially diagnosed neuroendocrine or small-cell carcinoma.
* Subjects with metastatic castration-resistant prostate cancer (mCRPC) who have failed novel androgen-deprived therapy and docetaxel chemotherapy. The previous antitumor treatment is ≥4 weeks prior to first dose.
* The previous clinical trials is ≥30 days prior to screening; Under the circumstance of previous clinical trials≤3 months , the pre-trial drug cannot interfere the safety and efficacy of current trial judged by the investigators.
* Age ≥18 years old when signing ICF, male, weight ≥50kg.
* Screening ECOG performance status is ≤2.
* Written information consent provided prior to the initiation of study procedures with cooperation during the follow-up.

Exclusion Criteria:

* Treatment requirement of Olaparib with the confirmed BRCA gene mutation.
* Rechallenge of docetaxel or other chemotherapy.
* Imminent Radiotherapy with radium-223.
* Plan to participate in other clinical trials.
* Pathological long bone fracture (cortical erosion > 50% on imaging) or spinal cord compression.
* History of other malignancies in the past 5 years with the exception of the following：cancer disease free≥5 years or squamous or basal cell skin carcinoma.
* Systemic therapy of immunosuppressive agents (such as cyclosporine, tacrolimus, rapamycin, and azathioprine, etc.) within one month prior to screening.
* Use of oral, intramuscular or intravenous corticosteroids within 28 days prior to enrollment. Short-term use of corticosteroids are allowed to prevent reactions for imaging studies. Use of inhaled corticosteroids for breathing insufficiency (chronic obstructive pulmonary disease) and topical steroids are allowed.
* Positive infectious disease screening. Active HBV hepatitis (defined as positive HBsAg with HBV-DNA ≥ upper limit of normal （ULN））; Active hepatitis C (defined as HBV-Ab ≥ULN)； Positive COVID-19；Human immunodeficiency virus (HIV) infection with HIV-Ab ≥ULN；Positive syphilis with TP-Ab≥ULN.
* Myocardial infarction, unstable angina pectoris, cardiac surgery or interventional therapy within 6 months prior to enrollment. Congestive heart failure, atrial fibrillation or other poorly controlled arrhythmias.
* Cerebrovascular events (including hemorrhagic, ischemic, transient ischemic attack), craniocerebral surgery and unexplained loss of consciousness occurred within 6 months before enrollment.
* Presence of the malignant pleural effusion or malignant ascites.
* History of severe allergic reactions or allergies to the ingredients of Prodencel.
* Abnormal screening hematologic function: white blood cell count (WBC)<3.0×109/L, neutrophil count (NEUT)<1.5×10^9/L, platelet count (PLT)<100×10^9/L, hemoglobin (Hb)< 100g/L.
* Abnormal screening coagulation function: prothrombin time (PT) ≥ULN, international normalized ratio (INR) ≥ULN, thrombin time (TT) ≥ULN.
* Abnormal screening liver and kidney function: total bilirubin (TBIL) > 1.5ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5ULN; serum creatinine (SCr) > 1.5 ULN.
* History of splenectomy.
* Presence of primary or secondary immunodeficiency disease.
* History of uncontrolled seizures, central nervous system disorders, or psychotic loss of cognition.
* History of chronic alcohol or drug abuse within 6 months prior to screening.
* Unstable systemic diseases, such as active infection, liver cirrhosis, chronic renal failure, severe chronic lung diseases, etc.
* Clinically severe pericardial effusion.
* Not suitable for leukapheresis.
* For any other reasons, the patients are believed not suitable for participation in this study by investigators.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs) during Induction Immunization | Up to 2 weeks after the third administration
  AEs were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs) during Booster Immunization | Up to approximately 1 year
  AEs were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Linhui Wang, Ph.D., Principal Investigator — Shanghai Changhai Hospital,The First Affiliated Hospital of Naval Medical University
Locations (1):
- Shanghai Changhai Hospital, The First Affiliated Hospital of Naval Medical University, Shanghai, Shanghai Municipality, China